CLINICAL TRIAL: NCT06143267
Title: Neuronostatin - a Glucagonotropic Agent in Humans?
Acronym: NSTCLAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Principal Investigator, Asger Lund, MD, MD, University Hospital, Gentofte, Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NSTCLAMP
Record Dates: First submitted 2023-11-09; First posted 2023-11-22 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes; Hypoglycemia; Type1diabetes
Keywords: Gut hormones; Alpha cell; Pancreas; Incretins
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, single-arm study. Each participant goes through six experimental days in a randomized order - acting as their own controls
Masking Description: The randomized order of infusions is blinded to both participant and investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Infusion of NST or placebo at different blood glucose levels (Experimental): In a randomized, double-blind crossover design, participants will undergo six experimental days with controlled plasma glucose levels, consisting of two euglycemic, two hyperglycemic (around 8mmol/l), and two hypoglycemic (around 2.5mmol/l) days, with each pair of similar days involving the administration of either saline (placebo) or NST.
  Interventions: Other: Infusion of either NST or placebo at different blood glucose levels

INTERVENTIONS:
Other: Infusion of either NST or placebo at different blood glucose levels — In a randomized, double-blind crossover design, participants will undergo six experimental days with controlled plasma glucose levels, consisting of two euglycemic, two hyperglycemic (around 8mmol/l), and two hypoglycemic (around 2.5mmol/l) days, with each pair of similar days involving the administration of either saline (placebo) or NST.

SUMMARY:
With the present study the investigators wish to delineate the effects of neuronostatin-13 (NST) on glucose-dependent glucagon secretion in humans. The main question it aims to answer is:

• What are the physiological effects of the naturally occuring hormone NST - especially with regards to glucagonotropic effects at different plasma glucose concentrations

In a randomized, double-blind crossover design, participants will undergo six experimental days with controlled plasma glucose levels, consisting of two euglycemic, two hyperglycemic (around 8mmol/l), and two hypoglycemic (around 2.5mmol/l) days, with each pair of similar days involving the administration of either saline (placebo) or NST.

DETAILED DESCRIPTION:
With the present study the investigators wish to delineate the effects of neuronostatin on glucose-dependent glucagon secretion in humans. Thus, this study is designed to elucidate the physiological effects of the natural occurring hormone, neuronostatin, and not to examine a medical effect of a drug or treatment. However, if neuronostatin acts glucagonotropically during low plasma glucose concentrations it could potentially help to address the unmet medical need for a treatment that, ultimately, can counteract the high risk of hypoglycaemia in patients treated with insulin.

After being informed about the study and the potential risks, each participant giving written informed consent will participate in six double-blinded experimental days (Day A-F) in a randomized order. On each day, participants will receive an infusion of either saline (placebo)(day A, C and E) or NST (day B, D and F). On day A and B, blood glucose will be kept at fasting levels, on day C and D blood glucose will be increased to ~8mmol/l and on day E and F blood glucose will be lowered to ~2.5mmol/l.

Blood glucose will be adjusted with insulin and/or glucose to reach the desired levels on each day.

At the end of the study day, participants will receive an ad libitum meal.

The effects of each infusion will be evaluated with regards to glucagonotropic potency, as well as a series of exploratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Normal haemoglobin >8.3 mmol/l
* Normal fasting plasma glucose below 7 mmol/l
* Normal HbA1C <42 mmol/mol (6%)
* Body mass index (BMI) 18.5-27 kg/m2
* Oral and written informed consent

Exclusion Criteria:

* Diabetes
* Treatment with drugs that might interfere with glucose metabolism within a month prior to the research study
* Treatment with any medication that cannot be paused for 12 hours
* Known liver disease and/or alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2 × normal values
* Nephropathy (eGFR <60 ml/min and/or albuminuria)
* Any condition that the investigator feels would interfere with trial participation

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Total glucagon response | 0-150minutes
  Differences in glucagon responses, measured as baseline subtracted AUC (bsAUC), between days with neuronostatin and placebo at corresponding glucose concentrations, respectively

SECONDARY OUTCOMES:
Glucagon response during first 60 minutes | 0-60minutes
  Differences in bsAUC for glucagon between days with neuronostatin and placebo at corresponding glucose concentrations, respectively, from 0 to 60minutes
Glucagon response during "recovery" | 60-90minutes
  Differences in bsAUC for glucagon between days with neuronostatin and placebo at corresponding glucose concentrations, respectively, from 60 to 90minutes
Glucagon response during hypoglycemia | t[BG=3.0] and the following 30 minutes
  Difference in bsAUC for glucagon between the two hypoglycemic study days with NST and placebo, respectively in the 30 minutes following a blood glucose (BG) below 3.0mmol/L
Total insulin response | 0-150minutes
  Difference in plasma levels of insulin between study days between days with neuronostatin and placebo at corresponding glucose concentrations, respectively
Total proinsulin-c-peptide response | 0-150minutes
  Difference in plasma levels of proinsulin-c-peptide between study days between days with neuronostatin and placebo at corresponding glucose concentrations, respectively
Amount of glucose infused | 0-150minutes
  Difference in infusion rates for glucose between study days between days with neuronostatin and placebo, respectively, at both hyperglycemic and hypoglycemic days
Difference in epinephrine | 0-150minutes
  Difference in plasma levels of epinephrine between days with neuronostatin and placebo at corresponding glucose concentrations, respectively
Difference in norepinephrine | 0-150minutes
  Difference in plasma levels of norepinephrine between days with neuronostatin and placebo at corresponding glucose concentrations, respectively
Difference in cortisol | 0-150minutes
  Difference in plasma levels of cortisol between days with neuronostatin and placebo at corresponding glucose concentrations, respectively
Difference in growth hormone | 0-150minutes
  Difference in plasma levels of growth hormone between days with neuronostatin and placebo at corresponding glucose concentrations, respectively
Difference in Procollagen 1 Intact N-Terminal Propeptide (P1NP) | 0-150minutes
  Difference in plasma levels of P1NP between days with neuronostatin and placebo at corresponding glucose concentrations, respectively
Difference in osteocalcin | 0-150minutes
  Difference in plasma levels of osteocalcin between days with neuronostatin and placebo at corresponding glucose concentrations, respectively
Difference in carboxy-terminal collagen crosslinks (CTX) | 0-150minutes
  Difference in plasma levels of CTX between days with neuronostatin and placebo at corresponding glucose concentrations, respectively
Difference in blood pressure | 0-150minutes
  Difference in blood pressure between days with neuronostatin and placebo at corresponding glucose concentrations, respectively
Difference in heart rate | 0-150minutes
  Difference in heart rate between days with neuronostatin and placebo at corresponding glucose concentrations, respectively
Energy expenditure | At -20 minutes, at 30 minutes, and at 75 minutes
  Difference in energy expenditure (measured by indirect calorimetry measuring respiratory gas exchange) between days with neuronostatin and placebo at corresponding glucose concentrations, respectively
Appetite | At -5 minutes, 25 minutes, 60 minutes, 90 minutes, and 120minutes
  Difference in appetite (assessed by visual analogue scale) between days with neuronostatin and placebo at corresponding glucose concentrations, respectively
Food intake | At 125 minutes
  Difference in food intake (assessed by ad libitum meal) between days with neuronostatin and placebo at corresponding glucose concentrations, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All published data will be made available to other researchers upon reasonable request